CLINICAL TRIAL: NCT01864720
Title: A Stepped Care Model for the Wider Dissemination of Cognitive-Behavioural Therapy for Insomnia Among Cancer Patients : Efficacy and Cost-Effectiveness.
Brief Title: Stepped Care Model for the Wider Dissemination of Cognitive-Behavioural Therapy for Insomnia Among Cancer Patients
Acronym: Stepped Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Josée Savard, Researcher, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC103664
Record Dates: First submitted 2013-05-21; First posted 2013-05-30 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Insomnia
Keywords: stepped care model; insomnia; cancer; cognitive-behavioural therapy; self-help treatment; web-based intervention; non-inferiority design; cost-effectiveness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Professionally Administered CBT-I (Standard Care) (Active Comparator): Patients (n = 59) assigned to this group will receive 6 weekly sessions of cognitive-behavioral therapy for insomnia (CBT-I) of approximately 50 minutes, offered individually by a licensed psychologist with significant experience (at least 2 years) in the administration of CBT-I with cancer patients.
  Interventions: Behavioral: Professionally-administered cognitive-behavioral therapy for insomnia (CBT-I)
- Stepped Care CBT-I (Experimental): Patients having an ISI score > 7 but < 15 (n = 65), will all receive first a web-based CBT-I for six weeks. Each week, the patients will first have to read written information on the website, and then watch a video capsule (duration between 5 and 20 min each). Patients with an ISI score > 14 (n = 53) will receive six weekly sessions of CBT-I administered individually by a professional.
  Interventions: Behavioral: Professionally-administered cognitive-behavioral therapy for insomnia (CBT-I); Behavioral: Web-based cognitive-behavioral therapy for insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Professionally-administered cognitive-behavioral therapy for insomnia (CBT-I) — The treatment content will be the same whether it is administered by a professional or self-administered. This multimodal approach combines behavioural (i.e., stimulus control therapy, sleep restriction), cognitive (i.e., cognitive restructuring), and educational (i.e., sleep hygiene) strategies that are administered over a 6-week period.
Behavioral: Web-based cognitive-behavioral therapy for insomnia (CBT-I) — The treatment content will be the same whether it is administered by a professional or self-administered. Each week, the patients will first have to read written information on the website, and then watch a video capsule (duration between 5 and 20 min each). The treatment material will be identical to the video (DVD)-based CBT-I that we previously developed. Patients will complete their daily sleep diary electronically on the website and the content will be interactive. It will include the sending of automated emails to remind participants to complete the treatment tasks and encourage adherence, provision of tailored feedback (e.g., texts, charts) based on the information that they provide in their sleep diary, as well as quizzes with automated correction to reinforce patients' understanding of the content.
  Other Names: Self-administered
  Arms: Stepped Care CBT-I

SUMMARY:
Insomnia is very common in cancer patients. When left untreated, insomnia can lead to numerous serious consequences (e.g., psychological disorders) for the individual and significant costs for society (e.g., increased medical consultations). Cognitive-behavioural therapy (CBT), a form of psychotherapy, is now considered the treatment of choice for insomnia and its efficacy has been demonstrated in clinical studies conducted in cancer patients. Unfortunately, CBT for insomnia (CBT-I) is not widely accessible as only a few cancer clinics have mental health professionals formally trained in the administration of this treatment. Innovative models of treatment delivery are therefore needed to make sure that every cancer patient with insomnia receives the care he/she needs. A stepped care approach in which patients only receive the level of treatment that they need, beginning with a minimal, less costly, intervention followed by more intensive treatment if required, has shown some promises for other psychological disorders (e.g., depression). Although its relevance has been emphasized to make CBT-I more accessible, its utility has never been investigated. The main goal of this randomized non-inferiority study is to assess the efficacy and costeffectiveness of a stepped care CBT-I as compared with standard care. Our hypothesis is that a stepped care approach will not be statistically inferior in terms of efficacy as compared to usual care, while being much less costly (better cost-effectiveness ratio). Three hundred cancer patients (mixed cancer sites) with insomnia symptoms will be assigned to: (1) stepped care CBT-I (n = 118) or (2) standard care (n = 59), consisting of 6 weekly sessions administered individually by a professional.

ELIGIBILITY:
Inclusion Criteria:

* have received a diagnosis of non-metastatic cancer (any type) in the past -18 months
* to have an ISI score > 7
* to be aged between 18 and 75 years old
* to be readily able to read and understand French

Exclusion Criteria:

* having a life expectancy < 1 year
* having a severe psychiatric disorder (e.g., psychotic, substance use, severe depressive disorder)
* having severe cognitive impairments (e.g., diagnosis of Parkinson's disease, dementia, or Mini-Mental State Examination score < 24)
* having received a formal diagnosis for another sleep disorder (e.g., obstructive sleep apnea, periodic limb movement disorder)
* shift work in the past 3 months or in the next 12 months
* to have received a CBT for insomnia in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2013-09; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  total score
Change in sleep efficiency (SE) index (%) | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  total sleep time/total time spent in bed X 100 - from sleep diary

SECONDARY OUTCOMES:
Change in sleep onset latency (SOL) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  time to sleep after lights out - from sleep diary
Change in wake after sleep onset (WASO) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  summation of nocturnal awakenings - from sleep diary
Change in total wake time (TWT) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  summation of SOL, WASO, and early morning awakening - from sleep diary
Change in total sleep time (TST) - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  time in bed minus total wake time - from sleep diary
Change in hypnotic use - from sleep diary | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  use of sleep-promoting medications - from sleep diary
Change in sleep onset latency (SOL) - from actigraphy | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  time to sleep after lights out - from actigraphy
Change in wake after sleep onset (WASO) - from actigraphy | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  summation of nocturnal awakenings - from actigraphy
Change in total wake time (TWT) - from actigraphy | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  summation of SOL, WASO, and early morning awakening - from actigraphy
Change in total sleep time (TST) - from actigraphy | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  time in bed minus total wake time - from actigraphy
Change in sleep efficiency (SE) index (%) - from actigraphy | Pre-tx (at recruitment; T1), post-tx (6 weeks after; T2), 3-month FU (T3), 6-month FU (T4), 12-month FU (T5)
  ratio of total sleep time to the actual time spent in bed multiplied by 100

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche de L'Hôtel-Dieu de Québec, Québec, Canada

REFERENCES:
- [Background] Espie CA. "Stepped care": a health technology solution for delivering cognitive behavioral therapy as a first line insomnia treatment. Sleep. 2009 Dec;32(12):1549-58. doi: 10.1093/sleep/32.12.1549. PMID 20041590
- [Background] Espie CA, Fleming L, Cassidy J, Samuel L, Taylor LM, White CA, Douglas NJ, Engleman HM, Kelly HL, Paul J. Randomized controlled clinical effectiveness trial of cognitive behavior therapy compared with treatment as usual for persistent insomnia in patients with cancer. J Clin Oncol. 2008 Oct 1;26(28):4651-8. doi: 10.1200/JCO.2007.13.9006. Epub 2008 Jun 30. PMID 18591549
- [Background] Savard J, Simard S, Ivers H, Morin CM. Randomized study on the efficacy of cognitive-behavioral therapy for insomnia secondary to breast cancer, part I: Sleep and psychological effects. J Clin Oncol. 2005 Sep 1;23(25):6083-96. doi: 10.1200/JCO.2005.09.548. PMID 16135475
- [Derived] Garneau J, Savard J, Dang-Vu TT, Gouin JP. Predicting response to stepped-care cognitive behavioral therapy for insomnia using pre-treatment heart rate variability in cancer patients. Sleep Med. 2024 Sep;121:160-170. doi: 10.1016/j.sleep.2024.06.021. Epub 2024 Jun 26. PMID 38991424
- [Derived] Savard J, Ivers H, Savard MH, Morin CM, Caplette-Gingras A, Bouchard S, Lacroix G. Efficacy of a stepped care approach to deliver cognitive-behavioral therapy for insomnia in cancer patients: a noninferiority randomized controlled trial. Sleep. 2021 Nov 12;44(11):zsab166. doi: 10.1093/sleep/zsab166. PMID 34228123